CLINICAL TRIAL: NCT01854866
Title: Phase II Study of Tumor Cell-derived Microparticles Used as Vectors of Chemotherapeutic Drugs to Treat Malignant Ascites and Pleural Effusion
Brief Title: Safety and Effectiveness Study of Tumor Cell-derived Microparticles to Treat Malignant Ascites and Pleural Effusion
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Bo Huang, professor, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soundny Biotech
Record Dates: First submitted 2013-04-12; First posted 2013-05-16 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Malignant Pleural Effusion,; Malignant Ascites
Keywords: Pleural Effusion; ascites; Malignant
MeSH Terms: conditions — Pleural Effusion, Malignant; Pleural Effusion; Ascites

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug-packaging Microparticles (Experimental): Drug-packaging microparticles are perfused to the pleural or peritoneal cavity of patients with four times per week.
  Interventions: Other: Drug-packaging microparticles

INTERVENTIONS:
Other: Drug-packaging microparticles — Drug-packaging microparticles are perfused to the pleural or peritoneal cavity of patients with four times per week.

SUMMARY:
Malignant ascites and pleural effusion are common symptoms in patients with advanced cancer. Currently, the management of malignant ascites and pleural effusion is a considerable clinical challenge. The investigator hypothesized that tumor cell-derived microparticles packaging chemotherapeutic drugs might be a useful means to treat malignant ascites and pleural effusion. Thirty malignant ascites or pleural effusion patients will be recruited for Phase II clinical trials.

DETAILED DESCRIPTION:
Ascites or pleural effusion were first removed from patients. The patients were then locally injected with microparticles packaging chemotherapeutic drugs 4 times a week. The therapeutic effects and side effects were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of malignant ascites or malignant pleural effusion

Exclusion Criteria:

* Non-malignant ascites or pleural effusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Volume of Ascites or Pleural Effusion | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Bo Huang, Ph.D, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Hubei Provincial Traditional Chinese Medical Hospital, Wuhan, Hubei, China

REFERENCES:
- [Background] Tang K, Zhang Y, Zhang H, Xu P, Liu J, Ma J, Lv M, Li D, Katirai F, Shen GX, Zhang G, Feng ZH, Ye D, Huang B. Delivery of chemotherapeutic drugs in tumour cell-derived microparticles. Nat Commun. 2012;3:1282. doi: 10.1038/ncomms2282. PMID 23250412
- See also: Related information — http://www.ncbi.nlm.nih.gov/pubmed/23250412